CLINICAL TRIAL: NCT00309478
Title: A Randomized Phase III Study Comparing Cyclophosphamide + Methotrexate + Fluorouracil vs. Goserelin + Tamoxifen in Premenopausal, Hormone Receptor-positive, Lymph Node-positive or -Negative Patients
Brief Title: Randomized Study Comparing CMF and Goserelin + Tamoxifen in Premenopausal Receptor-positive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABCSG-5
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Early-stage Breast Cancer
Keywords: Cyclophosphamide; Methotrexate; Fluorouracil; Goserelin; Tamoxifen; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Methotrexate; Fluorouracil; Goserelin; Tamoxifen

ARMS (2):
- 2 (CMF scheme) (Experimental): 6 cycles CMF scheme (cyclophosphamide, methotrexate, fluorouracil)
  Interventions: Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Fluorouracil implant
- 1 (Nol + Zol) (Experimental): Zoladex (3 years) combined with Nolvadex (5 years)
  Interventions: Drug: Goserelin; Drug: Tamoxifen

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 600mg/m2
  Arms: 2 (CMF scheme)
Drug: Methotrexate — Methotrexate 40mg/m2
  Arms: 2 (CMF scheme)
Drug: Fluorouracil implant — Fluorouracil 600mg/m2
  Arms: 2 (CMF scheme)
Drug: Goserelin — Zoladex 3.6mg/28 days for 3 years
  Other Names: Zoladex
  Arms: 1 (Nol + Zol)
Drug: Tamoxifen — Nolvadex 20mg/day for 5 years
  Other Names: Nolvadex
  Arms: 1 (Nol + Zol)

SUMMARY:
Primarily, this clinical investigation compared the efficacy of cyclophosphamide + methotrexate + fluorouracil chemotherapy vs. goserelin + tamoxifen treatment in terms of prognosis (disease-free survival, overall survival) in premenopausal patients with potentially curative, operated hormone receptor-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal patients with histologically verified, lymph node-negative (pT1c-pT3) or lymph node-positive (pT1a-pT3) breast cancer
* Hormone receptor-positive status
* More than 6 histologically examined lymph nodes
* Laboratory parameters

  1. hematopoiesis: > 3500/µl leukocytes, > 100,000/µl thrombocytes
  2. renal function: creatinin < 1.5mg %
  3. hepatic function: GOT </= 2.5 x UNL
  4. bilirubin: < 1.5mg %
  5. metabolic parameters: Na, Ca, K in normal range, normal level of blood sugar
  6. blood coagulation: PZ > 60%
* Concluded healing process following surgery
* </= 4 weeks interval since surgery
* Informed consent

Exclusion Criteria:

* T4 carcinoma; inflammatory breast cancer, carcinoma in situ
* Simultaneous or sequential bilateral breast cancer
* Preoperative tumor-reducing radiotherapy or preoperative tumor-specific medical treatment
* Male patients
* Pregnancy or lactation
* Lacking compliance or understanding of the disease
* General contraindication against cytostatic treatment
* Serious concomitant disease preventing implementation of adjuvant therapy or regular follow-up
* Second carcinoma or status post second carcinoma (except for curatively treated squamous cell carcinoma of the skin or cervical carcinoma in situ)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1099 (Actual)
Dates: Start 1990-12 (Actual); Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Disease-free survival
Overall survival

SECONDARY OUTCOMES:
Toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Jakesz, MD, Principal Investigator — Austrian Breast & Colorectal Cancer Study Group

REFERENCES:
- See also: Related Info — http://www.abcsg.at